CLINICAL TRIAL: NCT02645721
Title: Internet Based Cognitive Behavior Treatment for Alcohol Use Disorders - a Randomized Controlled Trial
Brief Title: Internet Based Cognitive Behavior Treatment for Alcohol Use Disorders
Acronym: ICBT-AUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/2014-31
Record Dates: First submitted 2016-01-02; First posted 2016-01-05 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Alcohol Use Disorders
MeSH Terms: conditions — Alcoholism | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Extended self-help program with guidance (Experimental): The program is a comprehensive CBT program lasting 12 weeks, with as many modules. The modules are quite extensive. A guide with basic education in psychotherapy assists and counsels participants online.
  Interventions: Behavioral: Extended self-help program with guidance
- Briefer Self-help program, no guidance (Active Comparator): This self-help program also lasts 12 weeks but contains only 9 modules; a pause occurs during the final weeks of the program for self-testing of acquired skills. The modules are quite brief. Participants receive no guidance.
  Interventions: Behavioral: Briefer Self-help program, no guidance
- WL: Extended self-help program, choice of guidance intensity (Other): Participants will be put on a waiting list. After 12 weeks on the waiting list, participants will receive access the the extended self-help program used in the experimental arm. However, participants will be offered a choice between three guidance options of varying intensity: proactive guidance, reactive guidance (only at participant request) or no guidance.
  Interventions: Behavioral: WL: Extended self-help program, choice of guidance intensity

INTERVENTIONS:
Behavioral: Extended self-help program with guidance — See arm description for Experimental
  Other Names: ePlus with guidance
  Arms: Extended self-help program with guidance
Behavioral: Briefer Self-help program, no guidance — See arm description for Active Comparator
  Other Names: eChange
  Arms: Briefer Self-help program, no guidance
Behavioral: WL: Extended self-help program, choice of guidance intensity — See arm description for Waiting list.
  Other Names: ePlus with choice of guidance intensity
  Arms: WL: Extended self-help program, choice of guidance intensity

SUMMARY:
The purpose of this study is to determine whether extensive internet based cognitive behavior treatment program with guidance is a more effective method to treat individuals with alcohol use disorders than a briefer cognitive behavior treatment program without guidance.

DETAILED DESCRIPTION:
Two Internet based programs based on cognitive behavioral therapy and relapse prevention are evaluated among Internet help seekers, and compared to a waiting list. The design is a three armed randomized controlled trial, and outcomes are measured in terms of changes in alcohol consumption (mean consumption/week, number of heavy drinking days/week), problematic alcohol use, self efficacy, craving, as well as depression, anxiety and quality of life. In addition to this, the following instruments will be used as predictors: ASRS (ADHD), Hp5i (personality assessment). TIC-P, an instrument measuring cost effectiveness will also be used. Treatment Credibility and Adverse Events will also be assessed, the former once during the third week of treatment, and the latter once half way through treatment and once after treatment.

Primary hypothesis is that the more extended program with guidance (group 1) is more effective in reducing mean alcohol consumption and number of heavy drinking days compared to the briefer program with no guidance (group 2), as well as compared to a waiting list (group 3). A responder to treatment is defined as a participant drinking less than 9 (women)/ 14(men) glasses per week and no more than 3 (women)/4 (men) glasses per drinking day during that week.

A minimum of 169 participants will be recruited in two phases: first through an online screening and then through a diagnostic telephone assessment, where SCID will be used to diagnose Alcohol Use Disorders and MINI will be used to diagnose other psychiatric diagnoses. The telephone assessment and all guidance will be conducted by licensed psychologists or master students in psychology under supervision by licensed psychologists.

Included participants will be randomized into three groups:

Group 1: All participants in this group will have access to an extended cognitive behavioral treatment program and have access to a guide with basic training in psychotherapy (CBT) who assists and counsels the participant throughout the program.

Group 2: Participants in this group will have access to a briefer cognitive behavior treatment program with no access to a guide.

Group 3: Participants in this group will be placed on a waiting list for 12 weeks. Thereafter, they will be given access to the same extended cognitive behavior treatment program as Group 1; they will also be offered a possibility to choose between three guidance options: Choice 1: guide with intensive support, Choice 2: guide with support only at request, Choice 3: no guide.

Interim analyses will be undertaken in May 2016 by graduate students in Clinical psychology writing their MSc theses.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* access to the internet
* consumption of at least 9 (females)/14 (males) glasses of alcohol during the preceding week
* AUDIT ≥ 14 for females, ≥ 16 for men
* have an Alcohol Use Disorder according to the DSM-5 (i.e., at least 2 out of 11 criteria)

Exclusion Criteria:

* insufficient Swedish skills
* reading or writing difficulties, if it is to a degree that it will hamper the treatment
* concurrent other psychological treatment with a content resembling treatments in this study
* severe depression defined as a score of more than 30 on the MADRS-S
* suicide-risk defined as more than 4 points on the MADRS-S question 9, or based on the structured interview
* Drug use problems defined as ≥ 8 p on the DUDIT
* somatic or psychiatric disorders that are contraindicated for the treatment or impairs the ability to receive it (for example schizophrenia, bipolar disease, PTSD)
* has during the last 3 weeks begun medication for alcohol problems or other psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back | Screening; Changes before treatment, Post-treatment (12 weeks); and changes after 3-, 12-, and 24-months post-treatment
  Number of standard drinks during preceding week (using the Time Line Follow Back)
Time Line Follow Back | Screening; Changes before treatment, Post-treatment (12 weeks); and changes after 3-, 12-, and 24-months post-treatment
  Days of heavy drinking during preceding week (using the Time Line Follow Back)

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test | Screening, Post-treatment (12 weeks), 3-, 12-, and 24-months post-treatment
  assessement of alcohol use problems
Alcohol Abstinence Self Efficacy Scale | Screening, Post-treatment (12 weeks), 3-, 12-, and 24-months post-treatment
  instrument measuring self-efficacy
Penn Alcohol Craving Scale | Screening, Post-treatment (12 weeks), 3-, 12-, and 24-months post-treatment
  instrument measuring craving for alcohol
Montgomery Asberg Depression Rating Scale | Screening, Post-treatment (12 weeks), 3-, 12-, and 24-months post-treatment
  instrument measuring depression
Euro-QOL 5 D | Screening, Post-treatment (12 weeks), 3-, 12-, and 24-months post-treatment
  instrument measuring quality of life
Generalized Anxiety Disorder-7 | Screening, Post-treatment (12 weeks), 3-, 12-, and 24-months post-treatment
  instrument measuring anxiety
Trimbos and iMTA questionnaire on cCosts associated with Psychiatric illness (TiC-P) | Screening, 12 months, 24 months post-treatment
  Instrument measuring health care consumption and cost-effectiveness (Bouwmans et al., 2013
Self-report questionnnaire on satisfaction with internet treatment usability features | Post-treatment (12 weeks after before-treatment measure)
  This instrument contains 40 questions about satisfaction with various features of the internet-based treatment. Results will be analyzed on an aggregated group level. The questionnaire was constructed by the Internet psychiatry clinic in Stockholm.
Adult ADHD Self Report Scale (ASRS) | Screening
  Screening of ADHD symptoms to be used as predictor of treatment outcome
Health-relevant Personality traits from a Five-factor perspective (hp5i) | Screening
  Screening of personality traits to be used as predictor of treatment outcome
Adverse Events | Halfway through treatment (6 weeks after before-treatment measure) and post-treatment (12 weeks after before-treatment measure)
  Brief questionnaire with questions about any negative side effects of the treatment
Treatment Credibility Scale | 3 weeks after before-treatment measure
  Brief questionnaire about if the treatment this far is perceived as effective
SCID- section of Alcohol Use Disorders (adjusted to DSM5) | Screening interview, 12 and 24 months post-treatment
  Diagnostic interview via telephone, diagnostic criteria of Alcohol Use Disorders (this will be undertaken if resurces allow). This will be a masked assessment, the interviewer will not know which original group the participant was randomized to

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided